CLINICAL TRIAL: NCT04692779
Title: A Prospective Clinical Study to Explore the Mechanism of Patients' Response to Prone Positioning in ARDS Patients, Including COVID-19
Brief Title: A Prospective Clinical Study to Explore Response to Prone Positioning in ARDS Patients
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Tyler Weiss, Clinical Education Coordinator, Rush University Medical Center
Other Study IDs: ProneARDS
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Covid19; ARDS
Keywords: Prone positioning; Lung ultrasound
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intubated ARDS patients undergoing prone positioning: All intubated ARDS patients undergoing prone positioning will be assessed with LUS before and after prone positioning and before and after placing back in the supine position.
  Interventions: Other: Lung Ultrasound (LUS)

INTERVENTIONS:
Other: Lung Ultrasound (LUS) — Enrolled subjects will undergo LUS 1 hour before and 1 hour after prone positioning by a trained clinician and will be assessed using a LUS score based on LUS pattern. LUS will then be performed again 1 hour before supination (16 hours) and assessed by a LUS score. This process will be repeated on the first 3 prone sessions. Patients will be enrolled in the study for 4 weeks in order to observe patient outcomes.

SUMMARY:
The proposed study will be conducted to investigate the mechanism of patients' responses to prone positioning with coronavirus disease 2019 (COVID-19) acute respiratory distress syndrome (ARDS) and non-COVID-19 ARDS utilizing lung ultrasound.

DETAILED DESCRIPTION:
This is a prospective observational study of adult patients with coronavirus disease 2019 (COVID-19) acute respiratory distress syndrome (ARDS) and non-COVID-19 ARDS who are intubated, in the prone position and receiving mechanical ventilation in the intensive care units at Rush University Medical Center. In this study design, we will prospectively enroll subjects, who fulfill eligibility criteria, to investigate the mechanism of their responses to the first three prone positioning sessions, utilizing lung ultrasound (LUS). Inclusion criteria include: adult subjects 18 years and older with a diagnosis of ARDS, endotracheally intubated and receiving assisted mechanical ventilation, meet criteria for prone positioning (ratio of arterial oxygen tension to the fraction of inspired oxygen (PaO2/FiO2) of ≤ 150 mm Hg with ventilator parameters of positive end-expiratory pressure (PEEP) ≥ 10 cm H2O and FiO2 of .60, and order for prone positioning. Patients will be excluded from the study if they meet the following criteria: pregnant, tracheostomy, receiving extracorporeal membrane oxygenation (ECMO), palliative care, received prone positioning more than once during intubation in an outside hospital, or receive invasive ventilation in an outside hospital for more than 72 hours. Enrolled subjects will undergo LUS 1 hour before and 1 hour after prone positioning by a trained clinician and will be assessed using a LUS score based on LUS pattern. LUS will then be performed again 1 hour before supination (16 hours) and assessed by a LUS score. This process will be repeated on the first 3 prone sessions. Patients will be enrolled in the study for 4 weeks in order to observe patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects 18 years and older, diagnosis of ARDS
2. endotracheally intubated and receiving assisted mechanical ventilation
3. meet criteria for prone positioning: PaO2/FIO2 (P/F ratio) of ≤ 150 mm Hg with ventilator parameters of PEEP ≥ 10 cm H2O and FiO2 of .60
4. receive an order for prone positioning.

Exclusion Criteria:

1. Pregnant
2. Tracheostomy
3. Receiving ECMO
4. Palliative care
5. Receive prone positioning more than once during intubation in an outside hospital
6. Receive invasive ventilation in an outside hospital for more than 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated adults (18 years or older) with a diagnosis of ARDS receiving mechanical ventilation and meet criteria for prone positioning.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Oxygenation and Lung Ultrasound Score (LUS) | 10 months
  Patients' responses of oxygenation and lung ultrasound score (0 - 36 where 0 = normal lung aeration and 36 = most severe lung consolidation) to prone positioning in the first three prone positioning sessions for ARDS patients.

SECONDARY OUTCOMES:
COVID-19 ARDS vs non-COVID-19 ARDS | 10 months
  observed lung ultrasound score (0 - 36 where 0 = normal lung aeration and 36 = most severe lung consolidation) differences between patients who respond to prone positioning and those who do not respond among patients with COVID-19 ARDS and non-COVID-19 ARDS.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Weiss, MS, Principal Investigator — Rush University Medical Center; Jie Li, PhD, Study Chair — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arbelot C, Ferrari F, Bouhemad B, Rouby JJ. Lung ultrasound in acute respiratory distress syndrome and acute lung injury. Curr Opin Crit Care. 2008 Feb;14(1):70-4. doi: 10.1097/MCC.0b013e3282f43d05. PMID 18195629
- [Result] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Result] Bouhemad B, Zhang M, Lu Q, Rouby JJ. Clinical review: Bedside lung ultrasound in critical care practice. Crit Care. 2007;11(1):205. doi: 10.1186/cc5668. PMID 17316468
- [Result] Doerschug KC, Schmidt GA. Intensive care ultrasound: III. Lung and pleural ultrasound for the intensivist. Ann Am Thorac Soc. 2013 Dec;10(6):708-12. doi: 10.1513/AnnalsATS.201308-288OT. No abstract available. PMID 24364779
- [Result] Haddam M, Zieleskiewicz L, Perbet S, Baldovini A, Guervilly C, Arbelot C, Noel A, Vigne C, Hammad E, Antonini F, Lehingue S, Peytel E, Lu Q, Bouhemad B, Golmard JL, Langeron O, Martin C, Muller L, Rouby JJ, Constantin JM, Papazian L, Leone M; CAR'Echo Collaborative Network; AzuRea Collaborative Network. Lung ultrasonography for assessment of oxygenation response to prone position ventilation in ARDS. Intensive Care Med. 2016 Oct;42(10):1546-1556. doi: 10.1007/s00134-016-4411-7. Epub 2016 Jun 20. PMID 27324241
- [Result] Prat G, Guinard S, Bizien N, Nowak E, Tonnelier JM, Alavi Z, Renault A, Boles JM, L'Her E. Can lung ultrasonography predict prone positioning response in acute respiratory distress syndrome patients? J Crit Care. 2016 Apr;32:36-41. doi: 10.1016/j.jcrc.2015.12.015. Epub 2015 Dec 30. PMID 26806842
- [Result] Wang XT, Ding X, Zhang HM, Chen H, Su LX, Liu DW; Chinese Critical Ultrasound Study Group (CCUSG). Lung ultrasound can be used to predict the potential of prone positioning and assess prognosis in patients with acute respiratory distress syndrome. Crit Care. 2016 Nov 30;20(1):385. doi: 10.1186/s13054-016-1558-0. PMID 27899151
- [Result] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Result] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Result] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Result] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Result] Munshi L, Del Sorbo L, Adhikari NKJ, Hodgson CL, Wunsch H, Meade MO, Uleryk E, Mancebo J, Pesenti A, Ranieri VM, Fan E. Prone Position for Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S280-S288. doi: 10.1513/AnnalsATS.201704-343OT. PMID 29068269
- [Result] Marini JJ, Hurford WE. Should Early Prone Positioning Be a Standard of Care in ARDS With Refractory Hypoxemia? Wrong Question-Reply. Respir Care. 2016 Nov;61(11):1564-1565. doi: 10.4187/respcare.05288. No abstract available. PMID 27794087
- [Result] Scholten EL, Beitler JR, Prisk GK, Malhotra A. Treatment of ARDS With Prone Positioning. Chest. 2017 Jan;151(1):215-224. doi: 10.1016/j.chest.2016.06.032. Epub 2016 Jul 8. PMID 27400909
- [Result] Kallet RH. A Comprehensive Review of Prone Position in ARDS. Respir Care. 2015 Nov;60(11):1660-87. doi: 10.4187/respcare.04271. PMID 26493592
- [Result] Reilly JP, Calfee CS, Christie JD. Acute Respiratory Distress Syndrome Phenotypes. Semin Respir Crit Care Med. 2019 Feb;40(1):19-30. doi: 10.1055/s-0039-1684049. Epub 2019 May 6. PMID 31060085
- [Result] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Result] Robba C, Battaglini D, Ball L, Patroniti N, Loconte M, Brunetti I, Vena A, Giacobbe DR, Bassetti M, Rocco PRM, Pelosi P. Distinct phenotypes require distinct respiratory management strategies in severe COVID-19. Respir Physiol Neurobiol. 2020 Aug;279:103455. doi: 10.1016/j.resp.2020.103455. Epub 2020 May 11. PMID 32437877
- [Result] Weiss TT, Cerda F, Scott JB, Kaur R, Sungurlu S, Mirza SH, Alolaiwat AA, Kaur R, Augustynovich AE, Li J. Prone positioning for patients intubated for severe acute respiratory distress syndrome (ARDS) secondary to COVID-19: a retrospective observational cohort study. Br J Anaesth. 2021 Jan;126(1):48-55. doi: 10.1016/j.bja.2020.09.042. Epub 2020 Oct 10. PMID 33158500